CLINICAL TRIAL: NCT06797141
Title: Combined Effects of Vestibular Rehabilitation and Dual Task Training Exercises on Balance, Gait and Quality of Life in Patients With Vestibular Disorders
Brief Title: Combined Effects of Vestibular Rehabilitation With Dual Task Training in Vestibular Disorders
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0257
Record Dates: First submitted 2024-11-03; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Vestibular Function Disorder
Keywords: Vestibular Disorders; Vestibular Rehabilitation; Dual Task Exercises; Quality of Life; Gait
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation and Dual Task Training and Traditional Physical Therapy (Experimental): Group A will receive treatment session lasting for 1 hour including vestibular rehabilitation therapy for 30 minutes and Dual Task Training for 20 minutes along with routine physical therapy of 10 minutes. Treatment session will be supervised by physical therapist and will be given 5 days per week for 8 weeks
  Interventions: Other: Vestibular Rehabilitation and Dual task Training and Traditional Physical Therapy
- Vestibular Rehabilitation and Traditional Physical Therapy (Active Comparator): Group B will receive treatment session lasting for 1 hour including vestibular rehabilitation therapy for 40 minutes along with routine physical therapy of 20 minutes. Treatment session will be supervised by physical therapist and will be given 5 days per week for 8 weeks.
  Interventions: Other: Vestibular Rehabilitation and Traditional Physical Therapy

INTERVENTIONS:
Other: Vestibular Rehabilitation and Dual task Training and Traditional Physical Therapy — Group A will receive treatment session lasting for 1 hour including vestibular rehabilitation therapy for 30 minutes and Dual Task Training for 20 minutes along with routine physical therapy of 10 minutes. Treatment session will be given 5 days per week for 8 weeks. Patients will be instructed to perform 2 sets of 5 repetition each Gaze Stability exercises: Horizontal and Vertical Head movements keep their eyes fixed on a stationary target, Following a slowly moving target keeping head still Balance Exercises:Maintain balance while performing neck rotations and shifting their weight forward, backward, and side to side.Sit to stand on chair Gait Training: Walking at varying speeds, walking forwards and backwards, sideways walking, walk in circles, and walking with horizontal and vertical head movements Dual Task exercises comprising of primary and secondary tasks Conventional Cawthorne Cooksey exercises :Up and down eye and Head movements, pick up things from ground, Walk up and down
  Arms: Vestibular Rehabilitation and Dual Task Training and Traditional Physical Therapy
Other: Vestibular Rehabilitation and Traditional Physical Therapy — Group B will receive treatment session lasting for 1 hour including vestibular rehabilitation therapy for 40 minutes along with routine physical therapy of 20 minutes. Treatment session will be given 5 days per week for 8 weeks.
  Gaze Stability exercises: Horizontal and Vertical Head movements keep their eyes fixed on a stationary target, Following a slowly moving target keeping head still Balance Exercises:Maintain balance while performing neck rotations and shifting their weight forward, backward, and side to side.Sit to stand on chair Gait Training: Walking at varying speeds, walking forwards and backwards, sideways walking, walk in circles, and walking with horizontal and vertical head movements Conventional Cawthorne Cooksey exercises :Up and down eye and Head movements, pick up things from ground, Walk up and down
  Arms: Vestibular Rehabilitation and Traditional Physical Therapy

SUMMARY:
Patients with vestibular disorders often experience cognitive-motor interference which can adversely affect their motor performance, significantly impair daily functioning, increase instability, reducing quality of life and increasing the risk of falls. Vestibular rehabilitation is a well-established therapeutic approach for managing vestibular disorders in reducing symptoms and improving balance and mobility. Similarly, Dual Task Training improves cognitive-motor integration by enhancing both cognitive and motor functions and has shown promising results in other populations. This study is aimed to determine the combined effects of both interventions as it might provide a more comprehensive and effective treatment, ultimately improving patient outcomes and quality of life.

DETAILED DESCRIPTION:
In previous studies, vestibular rehabilitation is well-documented in enhancing balance, gait, reducing dizziness and improving quality of life through specific exercises aimed at improving vestibular function. Similarly, dual task training has shown promise in improving functional mobility and cognitive processing. However, no randomized control trial to date has systematically investigated the potential synergistic effects of these two interventions when applied together which leaves a critical gap in understanding whether the integration of dual task training into vestibular rehabilitation could yield superior outcomes for patients suffering from vestibular disorders. This research could provide valuable insights and potentially enhance therapeutic strategies for this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of dizziness for longer than 3 months
* Patients with history of at least 1 bout of dizziness per month
* Patients with history of at least 1 fall in previous 6 months
* Diagnosed Patients as having vestibular disorder by an otolaryngologist
* Mini Mental State Examination (MMSE) score greater than 24

Exclusion Criteria:

* Patients with Meniere disease and bilateral vestibular disorders
* Patients with central nervous system disorders, and psychiatric disorders
* Patients having visual impairment that could not be treated with lenses or glasses
* Dizziness not resulting from vestibular disorder or use of Medication for Dizziness
* Movement limitation due to orthopedic problems
* Those who were unable to sign informed consent form

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go test | 8 week
  The instrument is used to assess dynamic balance including pace, distance, mechanism of turn, type of chair and number of trials. The time required to perform this test is measured. If more than 12 sec is taken in the completion of this test then it indicates high risk of fall
Dynamic Gait Index | 8 week
  Dynamic Gait Index (DGI) contains eight items measured on 4-point ordinal scale (3: Normal, 2: Mild Impairment, 1: Moderate impairment, 0: Severe Impairment).
Vestibular Rehabilitation Benefit Questionnaire | 8 week
  The Vestibular Rehabilitation Benefit Questionnaire (VRBQ) is 22 items subjective tool used to evaluate vestibular symptoms and their impact on quality of life in vestibular disorders. It is categorized into 3 subscales Dizziness and anxiety, Motion-provoked dizziness and Quality of life. Its score interpretation indicates 0%: no deficit & 100%: significant deficit. Score above 0% signifies the presence of symptoms, loss of function, or reduced quality of life

SECONDARY OUTCOMES:
Dizziness Handicap Inventory | 8 week
  It is a 25 item self-reported tool used to assess the level of disability experienced by individuals with dizziness, vertigo, or imbalance. It evaluates the impact of dizziness on functional, emotional, and physical aspects of the individual's life. It takes only 10 minutes to complete this tool. Patients rate their perceived disability due to dizziness by responding to each question with "yes," "sometimes," or "no." The answers are scored as follows: "No" = 0 points, "Sometimes" = 2 points, and "Yes" = 4 points. A higher total score, out of a possible 100 points, indicates a greater level of perceived disability. Patients scoring over 10 points should be referred for further evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Jabeen, PhD, Principal Investigator — Riphah International University
Locations (1):
- Fatima Memorial Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi WY, Gold DR. Vestibular Disorders: Pearls and Pitfalls. Semin Neurol. 2019 Dec;39(6):761-774. doi: 10.1055/s-0039-1698752. Epub 2019 Dec 17. PMID 31847047
- [Background] Aedo-Sanchez C, Riquelme-Contreras P, Henriquez F, Aguilar-Vidal E. Vestibular dysfunction and its association with cognitive impairment and dementia. Front Neurosci. 2024 Mar 27;18:1304810. doi: 10.3389/fnins.2024.1304810. eCollection 2024. PMID 38601091
- [Background] Strupp M, Dlugaiczyk J, Ertl-Wagner BB, Rujescu D, Westhofen M, Dieterich M. Vestibular Disorders. Dtsch Arztebl Int. 2020 Apr 24;117(17):300-310. doi: 10.3238/arztebl.2020.0300. PMID 32530417
- [Background] Staab JP. Persistent Postural-Perceptual Dizziness. Semin Neurol. 2020 Feb;40(1):130-137. doi: 10.1055/s-0039-3402736. Epub 2020 Jan 14. PMID 31935771